CLINICAL TRIAL: NCT03496532
Title: Optimization of Parameters of Subthalamic Nucleus Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study stoped becaus it did not even start No willing from our colleagues
Sponsor: Colette Boex (Other)
Responsible Party: Sponsor-Investigator, Colette Boex, Principal investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-01832
Record Dates: First submitted 2018-03-14; First posted 2018-04-12 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Poisson Distribution

STUDY DESIGN:
Intervention Model Description: Different stimulation paradigm tested sequentially in every patient of the group
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulse generator change under sedation (Experimental): The efficacy of every set will be measured on induced changes in LFP recorded from the STN electrodes.LFP will be compared between before, during and right after each stimulation conditions. The stimulation order will be randomized. All other stimulation parameters will be the same (macrocontact with most beta-oscillations, 1 minute, 1.5mA) .
  Hence 4 sets of 1 minutes of STN stimulation will be performed, for:
  Symmetrical biphasic pulses versus standard pseudo monophasic pulses (study I; 2 sets).
  Pseudorandom uniform distribution stimulation paradigms versus pseudorandom Poisson distribution stimulation paradigms (study II: 2 sets).
  Interventions: Device: biphasic stimulation; Device: standard stimulation; Device: Uniform distribution; Device: Poisson distribution
- First pulse generator implantation under general an (Experimental): The depth of anesthesia will be documented, recording the BIS spectral analysis index. The difference in spectral amplitude density of LFP, in particular in beta band oscillations will be correlated with the depth of anesthesia as measured with the BIS index.
  Interventions: Device: Recordings of LFP oscillations

INTERVENTIONS:
Device: biphasic stimulation — Fixed 70Hz symmetrical biphasic pulses
  Arms: Pulse generator change under sedation
Device: standard stimulation — Fixed 70Hz pseudo-monophasic pulses
  Arms: Pulse generator change under sedation
Device: Uniform distribution — Uniform distribution 70Hz Biphasic pulses
  Arms: Pulse generator change under sedation
Device: Poisson distribution — Poisson distribution 70Hz Biphasic pulses
  Arms: Pulse generator change under sedation
Device: Recordings of LFP oscillations — Two minutes of recordings of LFP oscillations will be performed from the contacts of the implanted electrode.
  Recordings of the depth of anaesthesia (BIS) all along the measurements performed under general anaesthesia.The correlation between the depth of anaesthesia and the cerebral oscillations recorded at the site of subthalamic nucleus will be studied.
  Arms: First pulse generator implantation under general an

SUMMARY:
Deep brain stimulation of the subthalamic nucleus is an effective treatment for Parkinson's disease. The analysis of cerebral signals of the subthalamic nucleus by local field potentials, provides one of the main electrophysiological markers of the success of the stimulation. This marker can be used to evaluate new paradigms of stimulation. So far, little studied, the temporal characteristics of the stimulation are very important in the effectiveness of the stimulation of the subthalamic nucleus, in Parkinson's disease. The first objective (Study I) is to compare the effectiveness of the stimulation when it is applied with biphasic symmetrical pulses and when applied with the standard pulses applied so far.

The second objective (Study II) is to see if, by applying pseudo-random time intervals between each stimulation pulse, if it would be possible to improve the efficiency and to limit the side effects of the stimulation.

The third objective (Study III) is to evaluate the electrophysiological changes of the subthalamic nucleus caused by the general anesthesia, in the anticipation of the realization of the surgery of the stimulation of the subthalamic nucleus under general anesthesia.

DETAILED DESCRIPTION:
Study I and II: Patients who participate undergo pulse generator change under sedation. Four sets of stimulation parameters will be compared. The efficacy of every set will be measured on induced changes in LFP recorded from the STN electrodes. LFP will be compared between before, during and right after each stimulation conditions. The stimulation order will be randomized. All other stimulation parameters will be the same (macrocontact with most beta-oscillations, 1 minute, 1.5mA) .

Study III: Patients who participate undergo their first pulse generator implantation, performed under general anesthesia because of wire tunnelisation. The depth of anesthesia will be documented, recording the BIS spectral analysis index. The difference in spectral amplitude density of LFP, in particular in beta band oscillations will be correlated with the depth of anesthesia as measured with the BIS index at the time of 2 minutes recordings.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from Parkinson's disease, who must undergo surgery for the replacement of their neurostimulator (under sedation) or for the first positioning of it
* capacity of discernment
* informed signed consent

Exclusion Criteria:

* Health considerations in regard to adding 13' in surgery room (e.g. pain or incomfort).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

PRIMARY OUTCOMES:
Comparison of quantity of Beta oscillations after biphasic pulses vs standard monophasic pulses | 10 minutes per patient
  % of changes in the energy of Beta oscillations
Comparison of quantity of Beta oscillations after pseudo random (Poisson distribution) vs uniform distribution of pulse time intervals | 10 minutes per patient
  % of changes in the energy of Beta oscillations
Observe the evolution of Beta oscillations during deep anesthesia | 2 minutes per patient
  Energy of Beta oscillations

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Switzerland